CLINICAL TRIAL: NCT04427631
Title: Exploring Interventions for Children With Chronic Otitis Media With Effusion ('Glue Ear') When Services Are Reduced During Covid-19
Brief Title: Exploring Interventions for Glue Ear During Covid-19
Acronym: BIG-C
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cambridgeshire Community Services NHS Trust (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr. Tamsin Brown, Paediatrician and chief investigator, Cambridgeshire Community Services NHS Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 262816
Record Dates: First submitted 2020-06-03; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Hearing Impaired Children; Glue Ear; Hearing Loss, Conductive
Keywords: Covid; OME; Glue ear; Otitis Media with effusion; paediatric; hearing loss
MeSH Terms: conditions — Otitis Media with Effusion; Hearing Loss, Conductive; Hearing Loss

STUDY DESIGN:
Intervention Model Description: single arm study offering all children with glue ear currently waiting on grommet operation lists, an invitation to be involved in this research study for hearing support (bone conduction headphones, a microphone and an app which can be delivered remotely)
Masking Description: It is too difficult to blind the assessor in thsi instance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm study (Experimental): The family will complete questionnaires before and after each childs intervention. Therefore each child will act as their own control.
  Interventions: Device: Bone conduction headphones

INTERVENTIONS:
Device: Bone conduction headphones — Children will be offered hearing support with bone conduction headphones that can either be paired to a microphone or to a tablet/ phone/ computer to help children to hear. The Hear Glue Ear app is available for free to provide speech and language enrichment.
  Other Names: Hear Glue ear app (software application)

SUMMARY:
During the Coronavirus pandemic children's hearing services are closed or reduced and grommet operations are part of the lowest priority group. In the absence of management options, this research study aims to see if bone conduction headphones either paired (via bluetooth) to a microphone or an app will help children with a hearing loss during this period of waiting. The child's quality of life is measured with validated questionnaires The study is over 3 months, and delivered remotely, with the product being sent to the family home and support offered via telephone/ video consulattion.

DETAILED DESCRIPTION:
Hypothesis

Transmission of speech aided by a wireless bone-conduction headphone connected to a wireless Bluetooth microphone during the prolonged waiting time (during the coronavirus pandemic) for the insertion of grommets, as well as access to the Hear Glue Ear software application is an acceptable management strategy during the coronavirus period where other forms of treatment and support are not available or indefinitely delayed. Questionnaires intend to capture data regarding families perception of child quality of life and developmental outcomes with this intervention.

Aim To quantify the differences in speech, language, and quality of life outcome measures between a group of children aided with a bone-conduction headphone and Hearing Glue Ear app during the coronavirus pandemic where usual care has been delayed such as waiting for grommet insertion.

Participants A total of 20 children will be enrolled in the study. If drop outs occur, new participants will be invited to replace those who withdrew from the study.

Participant recruitment Children known to Cambridge Audiology Services and known to have a diagnosis of glue ear will be invited to take part in the study if they satisfy the inclusion criteria. Consent will be obtained from their parents and an age appropriate explanation given to the child with the chance for the child to sign an age- appropriate assent form.

Design The free Hear glue Ear software application will be referred to as 'the app' in this section.

A single arm design will be used. Participants will have a glue ear (Otitis Media with Effusion, OME) diagnosis made in the National Health Service Cambridge Audiology clinics. They will be given information and invited to take part in the study at a time convenient to them.

Participants in the Study will be sent the bone conduction headphones, microphone and details of how to download the free Hear Glue Ear app. A member of the research team will arrange a telephone/ video consultation to aid set up and use of the product set.

The parent/ carer will be asked to fill out a questionnaire about their child's listening, language and quality of life before and after using the product set.

The bone conduction headphones used in this study are currently on the market as a headphones used by people practising outdoor sports. It is a type of headphones designed for children and adults to listen to music and speech via bluetooth to a phone or device. It is not a medical device but has a Conformity marking of Europe (known as CE mark) for being used as a set of headphones for any member of the public.

Follow-up will be carried out after 3 months unless the family request more frequent support. A member of the research team will email or telephone or video- consult (depending on the preference of the family) after 3 months to see if the family used the Hear Glue Ear headphones and/ or app at home and gather feedback. Parents will be asked to complete questionnaires again at this point.

The patient's family 'general practitioner' doctor will be informed (with parental consent) if the child is involved in the research study. The child's inclusion in the research study should not affect or alter any usual medical care.

Follow up will also be possible when the child attends their next NHS hearing test appointment when services reopen after or during the coronavirus pandemic.

Timing of the study and practical aspects

1. Invitation to take part

   The children and their families will be given a pack containing:
   * Parent and child study information sheets. The family and the child will have the chance to ask initial questions about the study within the remote telephone/ video clinic appointment.
   * Consent form, which the family can be encouraged to complete and return by email.

   Quality of life questionnaire for children with Otitis Media known as OMQ14 Speech, language and listening questionnaire.

   Website address: http://hearglueear.wordpress.com (study details including copies of consent forms and questionnaires will be available on the website) and contact email:

   hearglueear@outlook.com (for the families to direct any queries).
2. Once the child has been recruited

   * The children and their family will be sent a bone conduction headphone, microphone and information on how to download the free Hear Glue Ear app.
   * Participant's personal and contact details, as well as a copy of their last audiology results will be assigned a code that will be used for data collection, and their personal data and contact details will be kept separately.
   * Participating families will have a remote telephone/ video appointment offered at the beginning of the study and 3 months after their involvement.
3. Three months after their first appointment All the children will be automatically followed up with another telephone/ video consultation.

The family will be encouraged to fill out the final questionnaires, which are the same validated questionnaires used at the beginning of the study (before the intervention) as well as a non- validated acceptability questionnaire.

A website with videos, support information, instructions, and useful materials was created for use of the participants: http://hearglueear.wordpress.com

ELIGIBILITY:
Inclusion Criteria:

* Age 3-11y
* English used as a main language (since app is only written in English)
* Glue ear with a hearing loss affecting at least 2 frequencies in at least one ear

Exclusion Criteria:

* age range outside the 3-11 y parameter
* normal hearing
* not using english as a main language

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2020-06-22 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
acceptability of management strategy, questionnaire | Acceptability will be measured on a Likert scale pre-assessment and the end of 3 months of using the intervention
  questionnaire based accpetability question. A higher acceptability score will be positive for the intervention.

SECONDARY OUTCOMES:
quality of life questionnaire OMQ-14 | Questionnaires at beginning of study (as a baseline assessment and after 3 months of using the intervention. The sc
  validated questionnaire assessing quality of life in children with glue ear. The questionnaire assess disease- related hearing difficulty and treatment-related improvements in hearing. Improved (lower) scores will indicate a more positive response from the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Peacock Children's centre. Brookfields Hospital, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised individual patient data could be shared with other researchers as long as all personal information and details of a patients individual condition are unidentifiable (since it is a small study)